CLINICAL TRIAL: NCT01053117
Title: Reducing Hemodialysis Catheter Use in in a Prevalent Hemodialysis Population; A Pilot Randomized Control Trial
Brief Title: Reducing Hemodialysis Catheter Use in Prevalent Hemodialysis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enrol patients
Sponsor: Dr. Lisa Miller (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Sponsor-Investigator, Dr. Lisa Miller, Dr. Lisa Miller, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2008:101
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Hemodialysis
Keywords: central venous catheter; arteriovenous fistula; hemodialysis; vascular access; dialysis
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protocolized approach (Experimental): Protocolized approach to convert catheter to arteriovenous fistula
  Interventions: Other: Protocolized approach to convert dialysis catheter to fistula
- Current Care Model (No Intervention)

INTERVENTIONS:
Other: Protocolized approach to convert dialysis catheter to fistula — This group will be assigned an algorithm protocol in efforts to convert the central venous catheter to an arteriovenous fistula. A case manager will be assigned to follow these patients and implement the protocol
  Arms: Protocolized approach

SUMMARY:
To determine if a protocolized approach to converting hemodialysis central venous catheters (CVC) to arteriovenous fistulae will improve rates of functioning AVF and decrease CVC use.

DETAILED DESCRIPTION:
In order to receive dialysis, patients require repeated access to their bloodstream. This access can be either via a central venous catheter (CVC) or a surgically created arteriovenous fistula (AVF) or graft (AVG). This is a pilot randomized control trial of prevalent hemodialysis patients with a central venous catheter (CVC), to determine if a systematic approach using an algorithm protocol to convert the CVC to an AVF (arteriovenous fistula) will improve rates of functioning AVF and decrease CVC use. The algorithm (intervention group) will be compared to current practice (control group), a non-standardized approach at the discretion of the caring nephrologist and/or surgeon.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Dialyzing with a CVC
* Receiving hemodialysis three times weekly for > 3 months

Exclusion Criteria:

* Awaiting peritoneal dialysis catheter insertion
* Scheduled living donor transplant
* Transient patients from out of province
* Expected transfer to satellite dialysis unit within 6 months
* Surgical plan for AVF (i.e. scheduled date)
* Documented lack of suitable vasculature for AVF
* Refusing AVF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The proportion of patients using a CVC in a prevalent hemodialysis population after the implementation of an algorithm protocol to convert the CVC to an AVF compared with patients who received current standard care. | 9 months

SECONDARY OUTCOMES:
The proportion of patients with a functioning AVF after the implementation of an algorithm protocol to convert the CVC to an AVF compared with patients who received current standard care. | 9 months
Proportion of patients with a maturing AVF | 9 months
Primary fistula failure rate | 9 months
Incidence of AVF salvage procedures, including balloon angioplasty and accessory vein ligation, within 9 months of AVF creation | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Miller, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada